CLINICAL TRIAL: NCT06450132
Title: Longitudinal Changes in Eye Shape in Young Adults Treated With Low-Dose Atropine and Soft Multifocal Contact Lenses
Brief Title: Changes in Eye Shape With Myopia Management Interventions
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Donald O Mutti, OD, PhD, EF Wildermuth Foundation Professor in Optometry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023H0321
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The participants and the examining investigator will not be masked to intervention. All measurements are objective in nature and not subject to examiner bias. All data images acquired will be coded to obscure participant ID by a study team member masked to intervention. This coding will allow for the examining investigator to complete image processing while masked to randomization assignment, thereby minimizing the chance of bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Observation (No Intervention): Participants randomized to the observation arm will receive no intervention.
- Low-dose atropine (Experimental): Participants randomized to low-dose atropine will instill one drop of 0.05% atropine in each eye at bedtime for 12 months.
  Interventions: Drug: Atropine Ophthalmic
- Soft multifocal contact lenses (Experimental): Participants randomized to soft multifocal contact lenses will wear MiSight 1-day disposable contact lenses for 5-7 days per week for 12 months.
  Interventions: Device: MiSight 1-day disposable contact lenses

INTERVENTIONS:
Drug: Atropine Ophthalmic — 0.05% atropine ophthalmic solution
  Arms: Low-dose atropine
Device: MiSight 1-day disposable contact lenses — soft multifocal contact lenses
  Arms: Soft multifocal contact lenses

SUMMARY:
The goal of this clinical trial is to study changes in eye shape of nearsighted young adults using low-dose atropine eye drops or soft multifocal contact lenses. The main questions it aims to answer are:

* do low-dose atropine and soft multifocal contact lenses affect the shape of the peripheral eye?
* are changes in peripheral eye shape from these interventions influenced by changes in the focusing system of the eye?

Participants will:

* have multiple different types of photos taken
* have their prescription for glasses/contacts checked
* have their eye health checked, including the use of dilating eye drops
* be randomly assigned to use eye drops every night or wear special contact lenses daily instead of their typical contacts
* will complete five study visits over the course of 12 months

Researchers will compare young adults using low-dose atropine to those wearing soft multifocal contact lenses and to those using no intervention to see if using these interventions affects retinal shape.

ELIGIBILITY:
Inclusion Criteria:

* best corrected visual acuity of 20/25 or better in each eye
* nearsighted
* current contact lens wearer
* normal binocular vision (to be determined by an examiner at the first study visit)

Exclusion Criteria:

* eye diseases (including lazy eye or eye turn)
* pregnant, nursing, or planning a pregnancy in the next 12 months
* history of refractive surgery (e.g., LASIK)
* history of myopia control treatment
* sensitivity to anesthetics or preservative in eye drops
* difficulty with pupillary dilation

Ages: 21 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in ocular shape | baseline to 12 months
  ocular shape, as measured by the ellipsoid fit of the retina acquired by the photos taken with ocular ultrasound (ABSolu, Quantel Medical)

SECONDARY OUTCOMES:
Axial elongation (or regression) | baseline to 12 months
  change in axial length of the eye, as measured by Lenstar 900 (Haag-Streit)
Change in accommodative response | baseline to 12 months
  change in focusing ability of the eye, as measured with near targets and the Grand Seiko WR-5100K
Change in refractive error | baseline to 12 months
  change in refractive error, as measured with the Grand Seiko WR-5100K

CONTACTS AND LOCATIONS:
Overall Officials: Donald O Mutti, OD, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No